CLINICAL TRIAL: NCT03391817
Title: FAECAL MICROBIOTA TRANSPLANTATION IN THE TREATMENT OF MORBID OBESITY
Brief Title: FAECAL MICROBIOTA TRANSPLANTATION IN OBESITY
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Joint Authority for Päijät-Häme Social and Health Care (Other)
Collaborators: University of Helsinki (Other); Helsinki University Central Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FMTOBE
Record Dates: First submitted 2017-12-30; First posted 2018-01-05 (Actual); Last update posted 2019-08-15 (Actual); Status verified 2019-08

CONDITIONS: Obesity, Morbid
MeSH Terms: conditions — Obesity, Morbid | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Active Comparator): Fecal transplant from a thin donor
  Interventions: Other: Fecal microbiota transplantation
- Placebo arm (Placebo Comparator): Fecal transplant made from patients own feces
  Interventions: Other: Fecal microbiota transplantation

INTERVENTIONS:
Other: Fecal microbiota transplantation — Fecal microbiota transplantation administered in gastroscopy

SUMMARY:
40 patients meeting the criteria for obesity surgery are enrolled. Fecal microbiota transplantation (FMT) will be administered in gastroscopy 6 months before obesity surgery. 20 of the patients will receive a fecal transplant of a thin donor and 20 will receive placebo - a transplant made of their on feces. Changes in weight, laboratory values, general well being and stool microbiota will be measured up to one year after the surgery; one and a half years after FMT. The hypothesis is that FMT and the change in gut microbiota will help to reduce and maintain lower weight.

ELIGIBILITY:
Inclusion Criteria:

• Candidates for the bariatric surgery

BMI ≥ 40 or BMI ≥35 and at least two obesity-related co-morbidities such as type II diabetes (T2DM), hypertension, sleep apnea and other respiratory disorders, non-alcoholic fatty liver disease, osteoarthritis, lipid abnormalities, gastrointestinal disorders, or heart disease.

* Availability of consecutive fecal samples during one year
* Compliance to attend gastroscopy and FMT
* 18-65 years

Exclusion Criteria:

* Unable to provide informed consent
* Pregnancy
* Type I Diabetes Mellitus
* Severe renal insufficiency, GFR<30%
* Chronic or recurrent bacterial infection needing antimicrobial treatment
* Large hiatal hernia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-01-19 (Actual); Primary Completion 2021-02-28 (Estimated); Study Completion 2021-02-28 (Estimated)

PRIMARY OUTCOMES:
Reduction of weight | 1,5 years

CONTACTS AND LOCATIONS:
Overall Officials: Perttu Arkkila, PhD MD, Study Director — Helsinki University Central Hospital
Locations (2):
- Finland (2):
  - Helsinki University Hospital, Helsinki
  - Päijät-Häme Central Hospital, Lahti

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lahtinen P, Juuti A, Luostarinen M, Niskanen L, Liukkonen T, Tillonen J, Kossi J, Ilvesmaki V, Viljakka M, Satokari R, Arkkila P. Effectiveness of Fecal Microbiota Transplantation for Weight Loss in Patients With Obesity Undergoing Bariatric Surgery: A Randomized Clinical Trial. JAMA Netw Open. 2022 Dec 1;5(12):e2247226. doi: 10.1001/jamanetworkopen.2022.47226. PMID 36525272